CLINICAL TRIAL: NCT00982072
Title: Tacrolimus vs Prednisolone for the Treatment Minimal Change Disease
Brief Title: Tacrolimus Versus Prednisolone for the Treatment of Minimal Change Disease
Acronym: MinTAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13HH1283; 2009-014292-52 (EudraCT Number)
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Results first posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Minimal Change Disease
Keywords: nephrotic minimal change tacrolimus prednisolone
MeSH Terms: conditions — Nephrosis, Lipoid | interventions — Tacrolimus; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prednisolone (Active Comparator): prednisolone tablets
  Interventions: Drug: prednisolone
- tacrolimus (Experimental): tacrolimus tablets
  Interventions: Drug: tacrolimus

INTERVENTIONS:
Drug: tacrolimus — tacrolimus0.05mg/kg bd (levels 6-12ng/ml)
  Other Names: prograff
  Arms: tacrolimus
Drug: prednisolone — Prednisolone 1mg/kg maximum 60mg od
  Arms: prednisolone

SUMMARY:
The purpose of this study is to compare the effectiveness of tacrolimus (prograf) versus prednisolone for the treatment of nephrotic syndrome secondary to minimal change disease.

DETAILED DESCRIPTION:
Minimal change disease is a common cause of nephrotic syndrome in adults. Standard treatment is with high dose steroids which is often effective in controlling the nephrotic syndrome but has a high morbidity due to the side effects of the steroids. There is also a high relapse rate,therefore many patients require long term steroid therapy to control their disease which has significant morbidity and mortality. Some patients are or also become steroid resistant. There are studies showing the effectiveness of alkylating agents such as cyclophosphamide but the use of these drugs is limited by their toxicity, including increased rates of infection, cancers and infertility.

Tacrolimus (prograf) is a T-cell specific calcineurin inhibitor that shares similar immunosuppressive actions with cyclosporine A.In other glomerular diseases such as focal segmental glomerulosclerosis and membranous glomerulonephritis, prograf has been shown to be a very effective treatment for proteinuria. This may be due to the immunomodulatory effects on the underlying disease, but there may also be a direct effect of tacrolimus (prograf) on the podocyte, stabilising the actin cytoskeleton and therefore decreasing protein leak.Therefore tacrolimus (prograf) is likely to be effective in reducing proteinuria in minimal change disease.It has also been shown to have a good side effect profile when used to allow the avoidance of steroids in transplantation.This study aims to prospectively study if tacrolimus (prograf) is effective as treatment for minimal change disease compared with standard therapy with steroids, and whether it has advantages in terms of side effect profile and prevention of relapse.

ELIGIBILITY:
Inclusion Criteria:

* Patients with nephrotic syndrome (hypoalbuminaemia and protein creatinine ratio (PCR) > 100units), secondary to minimal change disease.
* Age over 18.

Exclusion Criteria:

* Hepatitis B, hepatitis C or HIV infection.
* Untreated infection.
* Females who are pregnant, breast feeding, or at risk of pregnancy and not using a medically acceptable form of contraception.
* Patients who have been treated with immunosuppression over the last 18 months.
* Patients who have had more than 3 relapses of nephrotic syndrome within 5 years.
* Any condition judged by the investigator that would cause the study to be detrimental to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Griffith, MBChBPhDFRCP, Study Chair — Imperial College NHS Trust; Tom Cairns, MBBSMRCP, Principal Investigator — Imperial College NHS Trust
Locations (1):
- Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Azukaitis K, Palmer SC, Strippoli GF, Hodson EM. Interventions for minimal change disease in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2022 Mar 1;3(3):CD001537. doi: 10.1002/14651858.CD001537.pub5. PMID 35230699

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prednisolone | Tacrolimus
Started | 25 | 27
Completed | 25 | 25
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prednisolone | Tacrolimus | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Customized [Count of Participants; unit: Participants]
  18 years and over | 25 | 27 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 15 | 25
  Male | 15 | 12 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 25 | 27 | 52

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Complete Remission From Nephrotic Syndrome at 8 Weeks
Description: normalisation of serum albumin and urine PCR <50 units
Time Frame: 8 weeks
Population: Patients at 8 weeks of therapy- on intention to treat basis
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisolone | Tacrolimus
Number analyzed (Participants) | 25 | 27
Participants | 21 | 17
Statistical Analysis 1: Comparison: Prednisolone vs Tacrolimus; Test type: Other; p = 0.12, Fisher Exact

2. Secondary Outcome: Percentage of Patients Achieving Complete Remission From Nephrotic Syndrome at 16 and 26 Weeks
Time Frame: 16 and 26 weeks
Population: Patients on intention to treat basis
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisolone | Tacrolimus
Number analyzed (Participants) | 25 | 27
Participants
  16 weeks | 23 | 19
  26 weeks | 23 | 22

3. Secondary Outcome: Percentage of Patients Achieving Remission Who Then Relapse
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisolone | Tacrolimus
Number analyzed (Participants) | 23 | 22
Participants | 17 | 16

4. Secondary Outcome: Number of Serious Adverse Events
Time Frame: 3 years
Measure: Number; unit: serious adverse events
Arm/Group | Prednisolone | Tacrolimus
Number analyzed (Participants) | 25 | 27
serious adverse events | 4 | 3

5. Secondary Outcome: Change in Baseline Glomerular Filtration Rate
Time Frame: 3 years
Population: data not collected
Arm/Group | Prednisolone | Tacrolimus
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Prednisolone | Tacrolimus
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/27
Serious Adverse Events (participants affected / at risk) | 4/25 | 3/27
Other Adverse Events (participants affected / at risk) | 18/25 | 20/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisolone (N=25) | Tacrolimus (N=27)
diverticualr disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 1 (1) | 0 (0)
fracture radius (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
hypertension (Cardiac disorders) | 0 (0) | 1 (1)
rash and diarhoaea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisolone (N=25) | Tacrolimus (N=27)
various non serious (General disorders) | 18 (18) | 20 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-02-02): https://cdn.clinicaltrials.gov/large-docs/72/NCT00982072/Prot_SAP_000.pdf